CLINICAL TRIAL: NCT00882739
Title: Safety and Efficacy of Three Different Loading Doses of Clopidogrel, Administered at First Medical Contact in Patients With Acute Myocardial Infarction Undergoing Primary Angioplasty. The LOAD & GO Trial
Brief Title: Safety and Efficacy of Three Different Loading Doses of Clopidogrel, in Patients With Acute Myocardial Infarction
Acronym: Load & Go
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Leonardo Bolognese, MD, Ospedale San Donato
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Arezzo002; EUDRACT 2009-010295-23
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Acute Myocardial Infarction
Keywords: angiography; percutaneous coronary intervention; Platelet Aggregation Inhibitors; Platelet Function Tests
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- no pre-treatment (Other): No pre-treatment at first medical contact - Patients will receive a 300 mg clopidogrel loading dose in the cath-lab setting
  Interventions: Drug: Clopidogrel 300 mg
- 600 mg loading dose (Experimental): 600 mg clopidogrel loading dose at first medical contact
  Interventions: Drug: Clopidogrel 600 mg
- 900 mg loading dose (Experimental): 900 mg clopidogrel loading dose at first medical contact
  Interventions: Drug: Clopidogrel 900 mg

INTERVENTIONS:
Drug: Clopidogrel 300 mg — Patients will receive a 300 mg clopidogrel loading dose in the cath-lab setting
  Other Names: Plavix-®
  Arms: no pre-treatment
Drug: Clopidogrel 600 mg — Patients will receive a 600 mg clopidogrel loading dose at first medical contact
  Other Names: Plavix-®
  Arms: 600 mg loading dose
Drug: Clopidogrel 900 mg — Patients will receive a 900 mg clopidogrel loading dose at first medical contact
  Other Names: Plavix-®
  Arms: 900 mg loading dose

SUMMARY:
The aim of this study is to determine both safety and effectiveness of three different loading dose regimens of clopidogrel in patients with acute myocardial infarction undergoing primary angioplasty.

DETAILED DESCRIPTION:
This study will enroll STEMI patients, who were planned to undergo PCI, and will randomize them to three different clopidogrel loading dose regimens at first medical contact: no pre-treatment, 600 mg or 900 mg. Platelet activity after administration of clopidogrel will be evaluated by VerifyNow™ P2Y12 point-of-care system.

The study is powered to demonstrate significant differences in the primary end point (the rate of TIMI Myocardial Perfusion Grade=3).

ELIGIBILITY:
Inclusion Criteria:

* ST-elevation myocardial infarction:

  * chest pain lasting more than 30 minutes
  * not responsive to nitrates
  * ST-segment elevation of more than 0.1 mV in two or more leads on the ECG, or new Left Bundle Branch Block
* With indication to primary PCI, presenting within 12 hour from symptoms onset
* Age > 18 years
* Planned PCI
* Informed Consent

Exclusion Criteria:

* bleeding diathesis
* allergy to study drugs
* pregnancy
* the performance of a rescue PCI after thrombolysis
* known existence of a disease resulting in a life expectancy of <6 months
* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
TIMI Myocardial Perfusion Grade (TMPG) | post-PCI

SECONDARY OUTCOMES:
TIMI flow | pre- and post-PCI
Corrected TIMI Frame Count (cTFC) | post-PCI
Major bleedings | 30 days
Major adverse cardiac events (MACEs) | 30 days
Platelet Reactive Units (PRU) as assessed by VerifyNow™ System | pre-PCI
TIMI 2-3 grade flow of the infarct-related artery | pre-PCI
no reflow phenomenon | post-PCI

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Bolognese, MD, FESC, Principal Investigator — Ospedale San Donato; Kenneth Ducci, MD, Principal Investigator — Ospedale San Donato
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy